CLINICAL TRIAL: NCT03918720
Title: In-depth Exploration of a Bidirectional Parent-child Health Relationship and Its Mediating Factors Among Low-income Families in Hong Kong
Brief Title: The Health and Effect of Health Empowerment Programmes Among Families in Tung Chung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Danny D B Ho Professor in Family Medicine and Department Head, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UW 12-517
Record Dates: First submitted 2017-11-03; First posted 2019-04-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Quality of Life; Empowerment
Keywords: Quality of Life; Empowerment; Low-income Families; Parent-child health relationship
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trekkers (Experimental)
  Interventions: Behavioral: Trekkers Family Health Empowerment Programme
- Controls (No Intervention)

INTERVENTIONS:
Behavioral: Trekkers Family Health Empowerment Programme — Health Assessment, Health Enablement and Health Literacy provided to empower participants awareness towards a healthier life style
  Other Names: Trekkers Family
  Arms: Trekkers

SUMMARY:
Kerry Group Kuok Foundation Limited (KGKF) has initiated the Trekkers Family Project that aims to enable low-income families to develop their full potentials by providing support and opportunities in education, employment, environmental harmony and health. Health is an essential component to enable a person to develop his/her full potential. This study looks into one of the key elements, health, of members of low-income families and the effect of health education, health enablement and mutual health support on health and social outcomes. It is a cohort study of around 800 subjects from 200 families of the Trekkers Family Project, and around 800 subjects not included in the Trekkers Family Project in Hong Kong, recruited base on pre-defined inclusion criteria. Health empowerment interventions consisting of three inter-related programmes, namely, the Health Literacy, the Self-care Enablement, and the Health Ambassador Programmes.

DETAILED DESCRIPTION:
The Health Literacy Programme aims to improve the knowledge on health and health services in order to promote health, prevent disease, and the proper use of services. It consists of four seminars per year on common health problems, mental health and cognitive health, etc.

The Self-Care Enablement Programme is to enable participants to keep themselves healthy, to build up self-efficacy and proper help-seeking skills, and to generate a spirit of mutual support among families. Two programmes will be delivered yearly, each with six 2.5 hour workshops facilitated by professional and lay leaders.

The Health Ambassador Programme aims to train up a group of adults recruited from the Trekkers families to act as a lay-advisor to other families on health issues. Participants who have completed the Health Literacy and Self-care Enablement programme will be given priority to take part in the Health Ambassador training programme.

The outcome measures are health enablement, health status, health-related quality of life, life style, cardiovascular risk factors, illnesses rates, and health service utilization pattern. All subjects in the cohort study will be surveyed on enrolment, and then yearly for 5 years. An age-gender appropriate health assessment will be carried out at baseline and at the end of five years for each subject. Changes in the outcomes will be evaluated and compared between groups. The impact of the health intervention programmes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Intervention group (inclusion criteria of Trekkers Families)

   1. Participants included must be part of a family whom all family members are usual residents in Tung Chung;
   2. The family must have at least one family member working full-time or part-time;
   3. The family household income does not exceed 75% of monthly median income of Hong Kong;
   4. At least one child studying Primary 1,2 or 3 at the time of recruitment; and
   5. At least one adult family member must be willing to participate in the long-term follow up study.
   6. Only fathers, mothers and children aged 6 or above will be included in this study.
2. Control group

   1. Participants included must be part of a family whom all family members are usual residents in Hong Kong;
   2. The family household income does not exceed 75% of monthly median income of Hong Kong;
   3. At least one child studying Primary 1, 2 or 3 at the time of recruitment;
   4. Only fathers, mothers and children aged 6 or above will be included in this study.

Exclusion Criteria:

1. None of the family member was able to understand or communicate in Chinese language,
2. The family is receiving Comprehensive Social Security Assistance (CSSA),
3. Refuse to give consent.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Patient enablement measured by the Chinese (HK) Patient Enablement Instrument at 60 months | Up to 60 months
  Patient Enablement Instrument-version 2 (PEI-2), score range 5 to 30, higher scores mean better enablement.

SECONDARY OUTCOMES:
Change from Baseline Health Status (global health, mental health) measured by DASS at 60 month | Up to 60 months
  Depression, Anxiety and Stress Scales (DASS), three subscales, each with a score range of 0 to 42, higher scores mean more emotional problems.
Change from Baseline Health-related quality of Life at 60 months | Up to 60 months
  12-item Short Form Health Survey-version 2 (SF-12v2) in adults: Physical Component Summary and Mental Component Summary scores, norm-based with a population mean of 50 and SD of 10, higher score means better quality of life.
  Child Health Questionnaire-Parent Form-28 items: Total Difficulty summary score ranges from 0-40, higher scores mean more behavioral difficulties; a prosocial scale score ranges from 0 to 10, higher scores mean better behavior.
Change from Baseline Lifestyle to 60 months | Up to 60 months
  proportion of participants with unhealthy lifestyle including smoking, <150min/wk of exercises, consumption of surgery drinks, smoking cigarettes, consumption of less than 5 portions of fruits and vegetables.
Change from Baseline Health parameters to 60 months | Up to 60 months
  Cardiovascular Health Index (CVHI) measured by optimal blood pressure, body mass index, blood cholesterol, blood glucose, smoking status, physical activity, and fruit and vegetable intake, score ranges from 0 to 7, higher scores mean better CVH.
Change from Baseline Health service utilization pattern to 60 months | Up to 60 months
  Proportion of people who reported to Have a family doctor, self-care for an illness, use of Accident and Emergency service during an illness episode.

OTHER OUTCOMES:
Change from Baseline Health knowledge test to 60 months | Up to 1 year
  pre and post knowledge test after each health education course.
Overall satisfaction after program | Up to 1 year
  Proportion of participants who reported overall satisfaction with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Lo Kuen Lam, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HRQOL of people from low-income families — http://doi.org/10.1016/j.jval.2015.09.2872
- See also: Protocol — http://doi.org/10.1136/bmjopen-2015-010015
- See also: Correlation of HRQOL between mothers and children — http://doi.org/10.15212/FMCH.2016.0124
- See also: Effect of intimate partner abuse on behaviour and HRQOL of children — http://doi.org/10.1007/s11136-017-1664-8
- See also: Maternal chronic disease and HRQOL of children — http://doi.org/10.1007/s40271-018-0314-8
- See also: Mobile app on parent-child exercises improves physical activity in children — https://doi.org/10.1186/s12889-020-09655-9
- See also: Health empowerment program improves cardiovascular health — https://doi.org/10.1016/j.pec.2024.108240
- See also: Health empowerment program improves HRQOL and behaviour in children — https://doi.org/10.1186/s13034-024-00834-9